CLINICAL TRIAL: NCT02261532
Title: A Phase 1, OPEN-Label, Non-randomized, Pharmacokinetic Study of TAS-102 in Chinese Patients With Solid Tumors
Brief Title: A Phase I Study of TAS-102 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10040100
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Results first posted 2024-10-18 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102 — TAS-102 (35 mg/m2/dose) orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics of TAS-102 after single and multiple dose in Chinese patients with solid tumor.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, single group Phase 1 study of TAS-102, evaluating the pharmacokinetics, safety, and antitumor activity. Blood sampling will be performed during the first cycle (Day1 and Day 12) of therapy in all consenting patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has provided written informed consent prior to performance of any study procedure.
* 2. Has definitive histologically or cytologically confirmed advanced or metastatic solid tumor.
* 3. Is able to take medications orally.
* 4. Has adequate organ function (bone marrow, kidney and liver).
* 5. Has Eastern Cooperative Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* 1. Has received TAS-102.
* 2. Has suffered serious complications.
* 3. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies.
* 4. Has had prior gastrectomy.
* 5. Is a pregnant or lactating female or male who refused using birth control during the clinical trial period and within 6 months after discontinuation of study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taiho Pharmaceutical Co., Ltd selected site, Beijing, China

REFERENCES:
- [Derived] Wang X, Zhou J, Li Y, Ge Y, Zhou Y, Bai C, Shen L. Pharmacokinetics, Safety, and Preliminary Efficacy of Oral Trifluridine/Tipiracil in Chinese Patients with Solid Tumors: A Phase 1b, Open-Label Study. Clin Pharmacol. 2020 Apr 9;12:21-33. doi: 10.2147/CPAA.S232104. eCollection 2020. PMID 32308505

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS-102
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAS-102
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 56.0 [35 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  China | 15

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Plasma Concentration) of FTD
Time Frame: Multiple time points on Day 1 and Day 12 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TAS-102
Number analyzed (Participants) | 14
ng/mL
  Day 1 | 3019.49 (34.0)
  Day 12 | 3693.08 (21.7)

2. Primary Outcome: Tmax (Time to Reach Maximum Drug Concentration in Blood) of FTD
Time Frame: Multiple time points on Day 1 and Day 12 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | TAS-102
Number analyzed (Participants) | 14
hours
  Day 1 | 1.00 (58.7)
  Day 12 | 2.61 (36.2)

3. Primary Outcome: AUC0-t (Area Under the Plasma Concentration Versus Time Curve From Time 0 to Time (t) of the Last Quantifiable Concentration ) of FTD
Time Frame: Multiple time points on Day 1 and Day 12 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | TAS-102
Number analyzed (Participants) | 14
ng·hr/mL
  Day 1 | 7796.60 (19.1)
  Day 12 | 18181.34 (30.0)

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | TAS-102
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-102 (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Platelet count decreased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-102 (N=15)
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastric dilatation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Protein urine present (Investigations) | 1
Urine bilirubin increased (Investigations) | 1
Fatigue (General disorders) | 7
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 3
Erythropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No